CLINICAL TRIAL: NCT04517981
Title: A Cohort Study on the Outcome and Influencing Factors of High-risk Pregnant Women With Perinatal Depression in the Third Trimester
Brief Title: Cohort Study on the Outcome and Influencing Factors of Perinatal Depression
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Mental Health Center, Jingan District (Other)
Responsible Party: Principal Investigator, Haiping Hu, Ward Director, Shanghai Mental Health Center, Jingan District
Other Study IDs: wcqyyzaywqgwyf
Record Dates: First submitted 2020-08-14; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Perinatal Depression; Prognosis
MeSH Terms: interventions — Psychosocial Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Drug intervention: Antidepressant
  Interventions: Behavioral: Psychological intervention; Other: Comprehensive intervention
- Psychological intervention: Cognitive behavior therapy, sand table therapy
- Comprehensive intervention: Psychological intervention, community intervention combined with drug intervention
  Interventions: Behavioral: Psychological intervention

INTERVENTIONS:
Behavioral: Psychological intervention — Choose according to the wishes of the enrolled subjects and the results of the evaluation
  Groups: Comprehensive intervention; Drug intervention
Other: Comprehensive intervention — Choose according to the wishes of the enrolled subjects and the results of the evaluation
  Groups: Drug intervention

SUMMARY:
1. Research and follow-up of the course and outcome of high-risk pregnant women with perinatal depression in the third trimester;
2. Factors affecting the outcome of the disease;
3. Recurrence of PND in pregnancy again;
4. The influence of different intervention methods on the course of the disease.

DETAILED DESCRIPTION:
Research objectives

1. Research and follow-up of the course and outcome of high-risk pregnant women with perinatal depression in the third trimester;
2. Factors affecting the outcome of the disease;
3. Recurrence of PND in pregnancy again;
4. The influence of different intervention methods on the course of the disease. Research process: 1. The pregnant women who were filed at Xinhua Hospital and Tongji Hospital and were receiving perinatal care from July 2019 to December 2019 were evaluated in the third trimester of pregnancy using the General Situation Questionnaire, SSRS, PHQ-9, and GAD-7. Those with PHQ-9 score ≥ 5 or GAD ≥ 5 were classified as having symptoms of depression and anxiety, and those who were screened positive were included in the study cohort; 42 days postpartum, 3 months postpartum, 6 months postpartum, 12 months postpartum, 18 months postpartum , 24 months postpartum, use PHQ-9, GAD-7 scale, 6 quality of life questionnaires, and SSRS to evaluate the cohort. If the PHQ-9 score is greater than or equal to 5 or the GAD is greater than or equal to 5, the psychiatrist will perform a clinical examination based on DSM-IV to make a clinical diagnosis; the outcome of the cohort and the incidence and influencing factors; 2 . During the follow-up process, the cohort developed high-risk pregnant women with depression, anxiety symptoms and other perinatal depressive disorders during the follow-up process. Based on the WeChat platform, integrated general hospitals, psychological counseling centers, social families and other service resources were carried out throughout the prenatal and first delivery period. Intervention methods such as community intervention for perinatal depression that focus on the comprehensive "physiology, psychology, and society" of the whole process after the first childbirth. Pregnant women diagnosed with PND will be evaluated by a psychiatrist to determine the treatment plan, and follow-up will continue.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Pregnant women in the third trimester (after 32 weeks of gestation);
  2. Shanghai resident pregnant women (for follow-up after delivery);
  3. Be able to complete perinatal care and infant health checkups in the research hospital;
  4. Decide to give birth in the research hospital;
  5. Willing to participate in this research and sign an informed consent form;
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Fate | 2019.9.1-2022.2.1
  Progression of high-risk pregnant women with perinatal depression in the third trimester
Influencing factors | 2019.9.1-2022.2.1
  Influencing factors of disease progression
Impact of intervention | 2019.9.1-2022.2.1
  The influence of different intervention methods on the course of the disease

CONTACTS AND LOCATIONS:
Overall Officials: huhaiping hp hu, Principal Investigator — Superior
Locations (1):
- Jing'an District Mental Health Center, Shanghai, Jing'an District, China

IPD SHARING:
Plan to Share IPD: Undecided